CLINICAL TRIAL: NCT03931096
Title: Quality of Life Assessment of Children With Congenital Heart Disease Aged 5 to 7 Years : a Multicentre Controlled Cross-sectional Study
Brief Title: Quality of Life Assessment of Children With Congenital Heart Disease Aged 5 to 7 Years
Acronym: QoL-CHD-5-7
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Pediatric and Congenital Cardiology Department of Necker-enfant malades University Hospital, Paris, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0061
Record Dates: First submitted 2019-04-08; First posted 2019-04-30 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Congenital Heart Disease
Keywords: health related quality of life; congenital heart disease; pediatrics; cardiology; PedsQL 4.0; psychometric properties
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with congenital heart disease: Groupe 1: case: children with congenital heart disease aged 5 to 7 years.
  Interventions: Other: Quality of life questionnaire
- control children: Groupe 2: control children recruited in schools aged 5 to 7 years.
  Interventions: Other: Quality of life questionnaire

INTERVENTIONS:
Other: Quality of life questionnaire — Self and proxy PedsQL 4.0 questionnaires.
  Other Names: Quality of life questionnaire: Pediatric Quality of Life Inventory Version 4.0 (PedsQL 4.0).

SUMMARY:
Congenital heart diseases (CHD) are the firt cause of congenital malformations (8 for 1000 births). Since the 90's, great advances in prenatal diagnosis, pediatric cardiac surgery, intensive care, and cardiac catheterization have reduced morbidity and early mortality in this population. Prevalence of " GUCH ", grown-ups with congenital heart disease has thus been significantly increasing. Nowadays, quality of life (QoL) assessment of this population is in the foreground. Our team is a reference center in the management of patient with CHD, from the fetal period to adulthood. The investigators have been conducting a clinical research program on health related QoL in pediatric and congenital heart disease. The investigators thus demonstrated the link between cardiopulmonary fitness and QoL in children with CHD aged 8 to 18 years, the correlation between functional class and QoL in adults with CHD, and the impact of therapeutic education on QoL in children under anticoagulants. Currently, no controlled cross-sectional quality of life study assessment has been leaded in the youngest children with CHD. This present study therefore extends our work in younger children aged 5 to 7 years.

DETAILED DESCRIPTION:
248 patients will be enrolled in this study.

Patient from groups 1 is included during his annual medical check-up. Quality of life questionnaire and other examinations are performed during this site visit. Its is a part of his usual care. No supplementary visit, directly related to the research, are necessary. 2 sites will participate to the enrollment, belonging to the French national network for complex congenital heart diseases (M3C) .

Participants (healthy children) from groups 2 are included from schools.The prior agreement of the Ministry of National Education was obtained before any procedure related to this study. 3 schools will participate to the enrolment

ELIGIBILITY:
Inclusion criteria:

• Children with CHD (as defined in the ACC-CHD classification) aged 5 to 7 years or same aged school children.

Exclusion criteria:

* Other comorbidity affecting quality of life (polymalformative syndrome, extracardiac organ failure, neurodegenerative disease, severe genetic disease, psychomotor retardation).
* Surgical procedure during the last 6 months.
* Inability to understand the QoL questionnaire (parents and / or child): non-french speaker, severe intellectual disability.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Groups 1 : Children with congenital heart disease aged 5 to 7 years Groups 2 : Healthy children aged 5 to 7 years
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
score of the self QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) | 1 day
  Comparison of the total score of the self QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) between patients with CHD and control children recruited in schools, aged 5 to 7 years. The self QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed.

SECONDARY OUTCOMES:
score of proxy QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) | 1 day
  Comparison of the total score of proxy QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) between patients with CHD and schoolchildren aged 5 to 7 years. The proxy QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed
score by dimensions of self and proxy QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) | 1 day
  Comparison of score by dimensions of self and proxy QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) between patients with CHD and schoolchildren aged 5 to 7 years.The proxy QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order o get score by dimensions of scale we must sum the items scores over the number of items answered. If more than 50% of the items in the scale are missing, the scale scores should not be computed.
score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the type of the CHD using the ACC-CHD classification. | 1 day
  Comparison of score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the type of the CHD using the ACC-CHD classification. The QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed.
score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the severity of the CHD using the BETHESDA classification. | 1 day
  Comparison of score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the severity of the CHD using the BETHESDA classification. The QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed
score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the patient functional status using the Ross classification. | 1 day
  Comparison of score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the patient functional status using the Ross classification. The QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed
score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the prognostic classification of the CHD using Davey B.T classification. | 1 day
  Comparison of score of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) to the prognostic classification of the CHD using Davey B.T. The QoL questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the Scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed
impact of variables related to the patient and to the CHD on his quality of life with the scores of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) | 1 day
  Study of the association of the following variables related to the patient and to the CHD with the scores of QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) . Univariate end multivariate analysis will be performed. The variables are:
  * sex of the patient,
  * age at diagnosis of CHD (pre or post natal)
  * number of cardiac surgeries
  * type of cardiac surgery (thoracotomy or sternotomy)
  * number of cardiac catheterizations
  * type of medical treatment
  * left ventricular ejection fraction (LVEF)
  * the presence of pulmonary arterial hypertension
  * the presence of a mechanical valve
  * the presence of a pacemaker or defibrillator
  * the presence of hypertension of the right ventricle.
Psychometric properties of the QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) . | 1 day
  Evaluation of the psychometric properties of the QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) .The Pediatric Quality of Life Inventory Version 4.0 (PedsQLTM 4.0) is a questionnaire widely used in pediatric clinical trials. This questionnaire was translated and linguistically validated in French, but no complete psychometric validation for French children has been performed yet. Reliability and validity are considered the main measurement properties of such instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Abassi H, Huguet H, Picot MC, Vincenti M, Guillaumont S, Auer A, Werner O, De La Villeon G, Lavastre K, Gavotto A, Auquier P, Amedro P. Health-related quality of life in children with congenital heart disease aged 5 to 7 years: a multicentre controlled cross-sectional study. Health Qual Life Outcomes. 2020 Nov 12;18(1):366. doi: 10.1186/s12955-020-01615-6. PMID 33183312